CLINICAL TRIAL: NCT03586349
Title: Cultural Adaptation of Sedentary Behavior Questionnaire and Reliability, Validity Research of Turkish Version
Status: Completed | Type: Observational
Sponsor: Begum Kara Kaya (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Sponsor-Investigator, Begum Kara Kaya, Lecturer, Biruni University
Organization: Biruni University (Other)
Other Study IDs: Study
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Healthy Adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to adapt the Sedentary Behavior Questionnaire (SBQ) into the culture of Turkish and to work on the reliability and validity of it in healthy individuals between the ages of 18-64. The permission was obtained via mail from Dori Rosenberg, who is the developer of the questionnaire, for its Turkish adaptation. SPSS package programme will be used in the analysis,

DETAILED DESCRIPTION:
The aim of this study is to adapt the Sedentary Behavior Questionnaire (SBQ) into the culture of Turkish and to work on the reliability and validity of it in healthy individuals between the ages of 18-64. Original form has nine questions but Spanish version of it had eleven questions so the investigators will translate Spanish version of SBQ. At first step by using a forward-backward translation method, a translation and adaptation process will be performed. At second step the validation process will be performed in a total of 200 healthy subjects aged between 18-64 years. Subjects will fill sociodemographic information form, International Physical Activity Questionnaire Short Form, and SBQ Turkish version ( at baseline and after seven days). Cronbach's alpha values, confirmatory factor analysis (CFA) will be evaluated for the reliability, construct and convergent validity.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy individual between the ages of 18-64.
* No problem of reading, writing or understanding Turkish.

Exclusion Criteria:

* Severe trauma in the last 6 months.
* Having orthopedic, neurological, cardiovascular problems that restricts ambulation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults aged between 18-64 years.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Sedentary Behavior Questionnaire | 1 week
  Sedentary Behavior Questionnaire scales the amount of time spent doing 11 sedentary behaviors.Response options are none, 15 minutes or less, 30 minutes, 1 hour, 2 hours,3 hours, 4 hours, 5 hours, 6 hours or more. In the scoring the time spent on each behavior is converted into hours (eg, a response of 15 minutes is recoded as .25 hours). For the total scores of sedentary behavior, responsed hours per day for each behavior are summed separately for weekday and weekend days. For the summary scores of total hours/day spent in sedentary behaviors (weekday and weekend) and total sedentary hours/week, responses higher than 24 hours/day are truncated to 24 hours/day. There are not any normative variables of Sedentary Behavior Questionnaire.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire Short Form | Day 1
  International Physical Activity Questionnaire Short Form(IPAQ-SF) scales the types of intensity of physical activity and sitting time that people do as part of their daily lives. The short form records the physical activity of 3 different intensity levels: 1) vigorous-intensity activity such as aerobics (8.0 MET), 2) moderate-intensity activity such as leisure cycling (4.0 MET), 3) walking (3.3 MET). The IPAQ-SF questions activities for last 7 days with 7 items. In the scoring total estimate physical activity in MET-min/week and time spent while sitting are calculated ( Ex. 4.0 METx activity dayx activity duration (in minutes) equals moderate-intensity activity total MET score).According to scores subjects are categorized as inactive (achieving <600 MET-min/week), minimally active (achieving a minimum of at least 600 MET-min/week and <3000 MET-min/week), active (>3000 MET-min/week).

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, Principal Investigator — Istanbul University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)